CLINICAL TRIAL: NCT04686422
Title: Clinical Evaluation of a Bulk Fill Resin Composite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LL3079573
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-04

CONDITIONS: Dental Caries; Unsatisfactory or Defective Restoration of Tooth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Tetric PowerFill Class I and II restorations (Experimental)
  Interventions: Device: Tetric PowerFill

INTERVENTIONS:
Device: Tetric PowerFill — Tooth (teeth) affected by dental caries or with an existing defective filling will be restored using the PowerCure system.

SUMMARY:
The purpose of this clinical trial is to measure the clinical outcomes of Tetric PowerFill Class I and II restorations cured in 3 seconds with the Bluephase PowerCure curing unit.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must need at least 1 restoration in a vital posterior tooth
* Must have given written consent to participate in the trial
* Replacement of defective restorations (i.e. fractured, stained, unaesthetic) with or with-out caries are acceptable
* Must be available for the required follow-up visits over 3 years
* Restored teeth must have occlusal contact with opposing teeth or restored teeth
* Restoration width should be equal to or greater than 1/3 the distance from buccal to lin-gual cusp tips
* 75% of the restorations Class II (minimum) and 25% Class I
* Each Class II will have at least one proximal contact
* 75% in molars (minimum) and 25% in premolars
* All restored teeth must have at least one occlusal contact in habitual closure
* Must have 20 or more teeth

Exclusion Criteria:

* If they have an allergy to ingredients of the materials under investigation (monomers)
* Do not meet all inclusion criteria above
* Have severe medical complications (organ transplants, long term antibiotic or steroid treatment, cancer or are immunocompromised) or disabilities meaning they may not be able to tolerate the time required to complete the restorations or to provide adequate oral hygiene
* Have xerostomia either by taking medications known to produce xerostomia or those with radiation-induced xerostomia or Sjogren's syndrome - as dry mouth increases tooth and restoration wear as well as the development of caries.
* Have teeth with advanced or severe periodontitis, rampant caries or poor oral hygiene which may require extraction of the teeth to be restored
* Present with any systemic or local disorders that contraindicate the dental procedures included in this study
* Have unstable occlusion
* Have severe grinding/bruxing or clenching or need TMJ-related therapy
* Have tooth with exposed pulp during preparation or caries removal
* Teeth that are non-vital or that exhibit signs of pulpal pathology for restoration
* Teeth that require cuspal build-ups involving more than one cusp

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Lawson, Dr, Principal Investigator — UAB School of Dentistry
Locations (1):
- UAB School of Dentistry, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Restorations
Period: Overall Study
Arm/Group | Tetric PowerFill Class I and II restorations
Started | 39; 68 Restorations
6 Month | 37; 66 Restorations
12 Month | 34; 62 Restorations
24 Month | 29; 52 Restorations
Completed | 23; 40 Restorations
Not Completed | 16; 28 Restorations

BASELINE CHARACTERISTICS:
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 39
Number analyzed (Restorations) | 68
Age, Customized [Count of Participants; unit: Participants]
  <= 18 years | 0
  Between 18 and 90 years | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0

OUTCOME MEASURES:

1. Primary Outcome: FDI 11 - Postoperative Hypersensitivity
Description: assessed by tests with thermal stimuli and occlusal forces (during biting) determined by VAS (Visual Analog Scale, 0 "No pain at all" - 10 "The worst pain imaginable") following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: Baseline
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 39
Number analyzed (Restorations) | 68
Restorations
  FDI Score 1 | 55
  FDI Score 2 | 10
  FDI Score 3 | 3
  FDI Score 4-5 | 0

2. Primary Outcome: Pulp Integrity
Description: Restored teeth are assessed by a cold air stimuli test (air syringe) by VAS (Visual Analog Scale, 0 "No pain at all" - 10 "The worst pain imaginable")
Time Frame: Baseline
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 39
Number analyzed (Restorations) | 68
Restorations
  VAS Score 0-1 | 60
  VAS Score 2-3 | 5
  VAS Score 4-6 | 2
  VAS Score 7-8 | 0
  VAS Score 9-10 | 1

3. Primary Outcome: Overall Survival Rate
Description: Restorations were examined by a dentist
Time Frame: Baseline
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 39
Number analyzed (Restorations) | 68
Restorations | 68

4. Primary Outcome: FDI 11 - Postoperative Hypersensitivity
Description: as for outcome 1
Time Frame: 6 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 37
Number analyzed (Restorations) | 66
Restorations
  FDI Score 1 | 60
  FDI Score 2 | 3
  FDI Score 3 | 3
  FDI Score 4-5 | 0

5. Primary Outcome: Pulp Integrity
Description: as for outcome 2
Time Frame: 6 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 37
Number analyzed (Restorations) | 66
Restorations
  VAS Score 0-1 | 64
  VAS Score 2-3 | 0
  VAS Score 4-6 | 0
  VAS Score 7-8 | 0
  VAS Score 9-10 | 2

6. Primary Outcome: Overall Survival Rate
Description: Restorations were examined by a dentist
Time Frame: 6 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 37
Number analyzed (Restorations) | 66
Restorations | 66

7. Primary Outcome: FDI 11 - Postoperative Hypersensitivity
Description: as for outcome 1
Time Frame: 12 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 34
Number analyzed (Restorations) | 62
Restorations
  FDI Score 1 | 59
  FDI Score 2 | 2
  FDI Score 3 | 1
  FDI Score 4-5 | 0

8. Primary Outcome: Pulp Integrity
Description: as for outcome 2
Time Frame: 12 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 34
Number analyzed (Restorations) | 62
Restorations
  VAS Score 0-1 | 60
  VAS Score 2-3 | 0
  VAS Score 4-6 | 2
  VAS Score 7-8 | 0
  VAS Score 9-10 | 0

9. Primary Outcome: Overall Survival Rate
Description: Restorations were examined by a dentist
Time Frame: 12 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 34
Number analyzed (Restorations) | 62
Restorations | 62

10. Primary Outcome: FDI 11 - Postoperative Hypersensitivity
Description: as for outcome 1
Time Frame: 24 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 29
Number analyzed (Restorations) | 52
Restorations
  FDI Score 1 | 50
  FDI Score 2 | 2
  FDI Score 3 | 0
  FDI Score 4-5 | 0

11. Primary Outcome: Pulp Integrity
Description: as for outcome 2
Time Frame: 24 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 29
Number analyzed (Restorations) | 52
Restorations
  VAS Score 0-1 | 49
  VAS Score 2-3 | 3
  VAS Score 4-6 | 0
  VAS Score 7-8 | 0
  VAS Score 9-10 | 0

12. Primary Outcome: Overall Survival Rate
Description: Restorations were examined by a dentist
Time Frame: 24 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 29
Number analyzed (Restorations) | 52
Restorations
  Survived | 51
  Failed | 1

13. Primary Outcome: FDI 11 - Postoperative Hypersensitivity
Description: as for outcome 1
Time Frame: 36 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 23
Number analyzed (Restorations) | 40
Restorations
  FDI Score 1 | 40
  FDI Score 2 | 0
  FDI Score 3 | 0
  FDI Score 4-5 | 0

14. Primary Outcome: Pulp Integrity
Description: as for outcome 2
Time Frame: 36 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 23
Number analyzed (Restorations) | 40
Restorations
  VAS Score 0-1 | 40
  VAS Score 2-3 | 0
  VAS Score 4-6 | 0
  VAS Score 7-8 | 0
  VAS Score 9-10 | 0

15. Primary Outcome: Overall Survival Rate
Description: Restorations were examined by a dentist
Time Frame: 36 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 23
Number analyzed (Restorations) | 40
Restorations
  Survived | 38
  Failed | 2

16. Secondary Outcome: FDI Criteria (Surface Lustre, Surface Staining, Colour Match, Material Fracture, Occlusal Wear, Tooth Integrity)
Description: assessed following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: Baseline
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 39
Number analyzed (Restorations) | 68
Restorations
  FDI 1 - Surface luster: FDI Score 1 | 68
  FDI 1 - Surface luster: FDI Score 2-5 | 0
  FDI 2 - Surface staining: FDI Score 1 | 68
  FDI 2 - Surface staining: FDI Score 2-5 | 0
  FDI 3 - Color matching: FDI Score 1 | 57
  FDI 3 - Color matching: FDI Score 2 | 8
  FDI 3 - Color matching: FDI Score 3 | 3
  FDI 3 - Color matching: FDI Score 4-5 | 0
  FDI 5 - Material fracture: FDI Score 1 | 68
  FDI 5 - Material fracture: FDI Score 2-5 | 0
  FDI 7 - Occlusal wear: FDI Score 1 | 68
  FDI 7 - Occlusal wear: FDI Score 2-5 | 0
  FDI 13 - Tooth integrity: FDI Score 1 | 68
  FDI 13 - Tooth integrity: FDI Score 2-5 | 0

17. Secondary Outcome: FDI Criteria (Surface Lustre, Surface Staining, Colour Match, Material Fracture, Occlusal Wear, Tooth Integrity)
Description: assessed following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: 6 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 37
Number analyzed (Restorations) | 66
Restorations
  FDI 1 - Surface luster: FDI Score 1 | 28
  FDI 1 - Surface luster: FDI Score 2 | 38
  FDI 1 - Surface luster: FDI Score 3-5 | 0
  FDI 2 - Surface staining: FDI Score 1 | 66
  FDI 2 - Surface staining: FDI Score 2-5 | 0
  FDI 3 - Color matching: FDI Score 1 | 61
  FDI 3 - Color matching: FDI Score 2 | 3
  FDI 3 - Color matching: FDI Score 3 | 2
  FDI 3 - Color matching: FDI Score 4-5 | 0
  FDI 5 - Material fracture: FDI Score 1 | 66
  FDI 5 - Material fracture: FDI Score 2-5 | 0
  FDI 7 - Occlusal wear: FDI Score 1 | 66
  FDI 7 - Occlusal wear: FDI Score 2-5 | 0
  FDI 13 - Tooth integrity: FDI Score 1 | 66
  FDI 13 - Tooth integrity: FDI Score 2-5 | 0

18. Secondary Outcome: FDI Criteria (Surface Lustre, Surface Staining, Colour Match, Material Fracture, Occlusal Wear, Tooth Integrity)
Description: assessed following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: 12 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 34
Number analyzed (Restorations) | 62
Restorations
  FDI 1 - Surface luster: FDI Score 1 | 25
  FDI 1 - Surface luster: FDI Score 2 | 37
  FDI 1 - Surface luster: FDI Score 3-5 | 0
  FDI 2 - Surface staining: FDI Score 1 | 59
  FDI 2 - Surface staining: FDI Score 2 | 3
  FDI 2 - Surface staining: FDI Score 3-5 | 0
  FDI 3 - Color matching: FDI Score 1 | 59
  FDI 3 - Color matching: FDI Score 2 | 3
  FDI 3 - Color matching: FDI Score 3 | 0
  FDI 3 - Color matching: FDI Score 4-5 | 0
  FDI 5 - Material fracture: FDI Score 1 | 62
  FDI 5 - Material fracture: FDI Score 2-5 | 0
  FDI 7 - Occlusal wear: FDI Score 1 | 62
  FDI 7 - Occlusal wear: FDI Score 2-5 | 0
  FDI 13 - Tooth integrity: FDI Score 1 | 62
  FDI 13 - Tooth integrity: FDI Score 2-5 | 0

19. Secondary Outcome: FDI Criteria (Surface Lustre, Surface Staining, Colour Match, Material Fracture, Occlusal Wear, Tooth Integrity)
Description: assessed following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: 24 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 29
Number analyzed (Restorations) | 52
Restorations
  FDI 1 - Surface luster: FDI Score 1 | 26
  FDI 1 - Surface luster: FDI Score 2 | 26
  FDI 1 - Surface luster: FDI Score 3-5 | 0
  FDI 2 - Surface staining: FDI Score 1 | 48
  FDI 2 - Surface staining: FDI Score 2 | 4
  FDI 2 - Surface staining: FDI Score 3-5 | 0
  FDI 3 - Color matching: FDI Score 1 | 51
  FDI 3 - Color matching: FDI Score 2 | 1
  FDI 3 - Color matching: FDI Score 3 | 0
  FDI 3 - Color matching: FDI Score 4-5 | 0
  FDI 5 - Material fracture: FDI Score 1 | 52
  FDI 5 - Material fracture: FDI Score 2-5 | 0
  FDI 7 - Occlusal wear: FDI Score 1 | 50
  FDI 7 - Occlusal wear: FDI Score 2 | 2
  FDI 7 - Occlusal wear: FDI Score 3-5 | 0
  FDI 13 - Tooth integrity: FDI Score 1 | 52
  FDI 13 - Tooth integrity: FDI Score 2-5 | 0

20. Secondary Outcome: FDI Criteria (Surface Lustre, Surface Staining, Colour Match, Material Fracture, Occlusal Wear, Tooth Integrity)
Description: assessed following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: 36 Month
Measure: Number; unit: Restorations
Units Other Than Participants: Restorations
Arm/Group | Tetric PowerFill Class I and II restorations
Number analyzed (Participants) | 23
Number analyzed (Restorations) | 40
Restorations
  FDI 1 - Surface luster: FDI Score 1 | 12
  FDI 1 - Surface luster: FDI Score 2 | 28
  FDI 1 - Surface luster: FDI Score 3-5 | 0
  FDI 2 - Surface staining: FDI Score 1 | 40
  FDI 2 - Surface staining: FDI Score 2-5 | 0
  FDI 3 - Color matching: FDI Score 1 | 35
  FDI 3 - Color matching: FDI Score 2 | 5
  FDI 3 - Color matching: FDI Score 3 | 0
  FDI 3 - Color matching: FDI Score 4-5 | 0
  FDI 5 - Material fracture: FDI Score 1 | 40
  FDI 5 - Material fracture: FDI Score 2-5 | 0
  FDI 7 - Occlusal wear: FDI Score 1 | 36
  FDI 7 - Occlusal wear: FDI Score 2 | 4
  FDI 7 - Occlusal wear: FDI Score 3-5 | 0
  FDI 13 - Tooth integrity: FDI Score 1 | 40
  FDI 13 - Tooth integrity: FDI Score 2-5 | 0

ADVERSE EVENTS:
Time Frame: 36 Months
Arm/Group | Tetric PowerFill Class I and II restorations
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 2/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tetric PowerFill Class I and II restorations (N=39)
Restoration was replaced (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT04686422/Prot_SAP_001.pdf